CLINICAL TRIAL: NCT00009958
Title: A Phase I Study of Sequential Vaccinations With Fowlpox-CEA(6D)-TRICOM (B7.1/ICAM/LFA-3) Alone, and in Combination With Vaccinia-CEA(6D)-TRICOM, and the Role of GM-CSF, in Patients With CEA Expressing Carcinomas
Brief Title: Vaccine Therapy With or Without Sargramostim in Treating Patients With Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03151; IBC20-09; P30CA051008 (NIH); NCI-833; NIH/OBA-0006-405; CDR0000068427; GUMC-IBC20-09; GUMC-00101
Record Dates: First submitted 2001-02-02; First posted 2004-02-03 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (3):
- Stage I (Experimental): Patients receive fCEA-TRI vaccine SC once daily on days 1, 29, 57, and 85.
  Interventions: Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Other: laboratory biomarker analysis
- Stage II (Experimental): Patients receive vCEA-TRI vaccine intradermally once on day 1 and fCEA-TRI vaccine SC at the MTD determined in stage I once daily on days 29, 57, and 85.
  Interventions: Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Biological: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Other: laboratory biomarker analysis
- Stage III (Experimental): A single cohort of 6-10 patients receive both vaccines as in stage II, at the MTDs determined in stages I and II, and sargramostim (GM-CSF) SC once daily on days 1-4, 29-32, 57-60, and 85-88.
  Interventions: Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Biological: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Biological: sargramostim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine — Given SC
  Other Names: fowlpox-CEA-B7-1/ICAM-1/LFA-3; rF-CEA(6D)TRICOM
Biological: recombinant vaccinia-CEA(6D)-TRICOM vaccine — Given intradermally
  Other Names: rV-CEA(6D)-TRICOM
  Arms: Stage II; Stage III
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
  Arms: Stage III
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to compare the effectiveness of vaccine therapy with or without sargramostim in treating patients who have solid tumors. Vaccines may make the body build an immune response to kill tumor cells. Combining colony-stimulating factors such as sargramostim with vaccines may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and toxicity profile of the novel CEA-based vaccine, rF-CEA(6D)-TRICOM (recombinant fowlpox-CEA(6D)-B7.1/ICAM-1/LFA-3), either alone or in combination with a second vaccine, rV-CEA(6D)-TRICOM (recombinant vaccinia-CEA(6D)-B7.1/ICAM-1/LFA-3) in patients with advanced CEA-bearing cancers.

II. To determine the maximum tolerated dose and toxicity profile of the novel CEA-based vaccine rV-CEA(6D)-TRICOM when given in combination with the maximum tolerated dose of rF-CEA(6D)-TRICOM, in patients with advanced CEA-bearing cancers.

III. To determine the safety and impact of colony stimulating factors (GM-CSF) on the immunologic response, when given in conjunction with the combination of rV-CEA(6D)-TRICOM (MTD) and rF-CEA(6D)-TRICOM (MTD) vaccines, in patients with advanced CEA-bearing cancers.

IV. To determine the change in CAP-1 directed T cells in patients treated with these vaccines using ELISPOT assay analysis.

V. To perform a pilot analysis of the impact of vaccine therapy on the quantity of circulating CEA-positive cells in the patients treated on this study in order to develop and eventually validate a practical, intermediate bio-marker for the immunologic response to the vaccines.

VI. To document any objective anti-tumor responses that occur.

OUTLINE: This is a dose-escalation study of fowlpox-CEA-TRICOM (fCEA-TRI) vaccine and vaccinia-CEA-TRICOM (vCEA-TRI) vaccine.

STAGE I: Patients receive fCEA-TRI vaccine subcutaneously (SC) once daily on days 1, 29, 57, and 85.

Cohorts of 3-10 patients receive escalating doses of the fCEA-TRI vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity (DLT).

STAGE II: Patients receive vCEA-TRI vaccine intradermally once on day 1 and fCEA-TRI vaccine SC at the MTD determined in stage I once daily on days 29, 57, and 85.

Cohorts of 3-10 patients receive escalating doses of the vCEA-TRI vaccine until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT.

STAGE III: A single cohort of 6-10 patients receive both vaccines as in stage II, at the MTDs determined in stages I and II, and sargramostim (GM-CSF) SC once daily on days 1-4, 29-32, 57-60, and 85-88.

Patients in any stage of the study with responding disease may receive additional doses of the fCEA-TRI vaccine monthly for 2 months and then every 3 months thereafter. Patients who have objective evidence of response (including mixed response) and/or a fall in an elevated serum CEA level after the sixth vaccine and who subsequently develop disease progression while on the extended every 3-month treatment schedule and have no other potentially better treatment alternatives available may continue treatment as per the monthly vaccination schedule for 2 additional months. Patients with stable or responding disease after those two monthly vaccines may continue monthly vaccines at the discretion of the principal investigator.

Patients are followed at 4 weeks and then monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of malignancy, with evidence of metastatic disease (evaluable disease is adequate), who have not responded to standard therapy, who have relapsed, or for whom such therapy is not available
* Patients must have a tumor that has been shown to express CEA by immunohistochemical techniques or have had an elevated serum CEA > 10 at any point during their disease course
* Patients must have an anticipated survival of at least 6 months
* Patients must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects), and must sign an informed consent
* Patients must be ambulatory, with an ECOG performance status of 0 or 1, and must be maintaining a reasonable state of nutrition, consistent with weight maintenance
* WBC >= 3,000/mm^3
* ANC >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin =< 2 x upper limit of normal
* SGOT and SGPT =< 4 x upper limit of normal
* All patients should have an initial urine analysis; the initial urine analysis for eligibility is: proteinuria grade 0, hematuria grade 0, and no abnormal sediment; any positive protein including trace values should be evaluated by a 24-hour urine; any other abnormality in the sediment or the presence of hematuria should be evaluated by a nephrologist for evidence of underlying renal pathology; patients may be eligible if the underlying cause of the abnormality is determined to be non-renal
* Normal creatinine is defined by creatinine =< 1.5 mg/dL OR creatinine clearance >= 60 ml/min
* At least 6 patients must be HLA-A2 positive for each of cohorts 3, 6, and 7; once the HLA-A2 positive quota of 6 has been met, enrollment to that cohort may close at the discretion of the principal investigator; there are no HLA phenotype restrictions for cohorts 1,2,4, and 5, although phenotyping will be performed on all patients
* Vaccinia-naïve patients may be enrolled to any cohort

  * There must be no history of allergy or untoward reaction to prior vaccination with vaccinia virus, for patients on cohorts 4, 5, 6, or 7
* Patients for all cohorts should have no evidence of immunocompromise or autoimmunity as defined by:

  * HIV negative by serologic testing; this requirement is due to the potential for an unacceptable high risk of systemic viremia, if live virus vaccine were to be administered to an immunocompromised individual; while similar constructs have been given to HIV positive patients, concern is high for toxicity, particularly with vaccinia
  * No other diagnosis (past or present) of:

    * Altered immune function, including immunodeficiency or history of immunodeficiency; eczema; history of eczema, or other eczematoid skin disorders; or those with acute, chronic or exfoliative skin conditions (e.g. atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds; this requirement is due to a potential unacceptable high risk of systemic viremia, if study vaccine were to be administered to an immunocompromised individual
    * Any autoimmune disease such as, Addison's disease, Hashimoto's thyroiditis, or systemic lupus erythematous, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome active Grave's disease; this requirement is due to the potential risks of autoimmunity
  * No prior radiation to > 50% of all nodal groups
  * No concurrent use of systemic steroids, except for physiologic doses for systemic steroid replacement or local (topical, nasal, or inhaled) steroid use
* Patients must have recovered from the reversible side effects of prior therapy
* Patients must be willing and able to travel to Georgetown University Hospital for treatment and follow-up during therapy and at least monthly thereafter until there is evidence of disease progression
* Patients must be able to avoid close household contact (close household contacts are those who share housing or have close physical contact) with persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children under 5 years of age; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV infection

Exclusion Criteria:

* Recent major surgery (within 21 days)
* Frequent vomiting or severe anorexia
* Pregnant or lactating women; this requirement is due to an unacceptable high risk of CEA antibody transfer, which may be potentially harmful to the developing fetus or infant; (NOTE: women and men enrolled in the study are to practice an effective method of birth control for at least six months after their last treatment on protocol)
* Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis
* The following therapies are prohibited and may not be administered to patients being treated on this protocol: chemotherapy, hormonal therapy, biologic therapy, and immunotherapy
* Patients must have recovered completely from any reversible toxicity associated with their most recent therapy; typically this is 3-4 weeks for patients who most recently received cytotoxic therapy except for the nitrosoureas and mitomycin C for which 6 weeks is needed for recovery
* Patients with clinically active brain metastasis, uncontrolled seizure disorders, encephalitis, or multiple sclerosis
* Patients can not have any history (past or present) of allergy to eggs or egg products
* Patients with history of receiving CEA-containing vaccines are excluded from enrollment into any of the 8 actual study cohorts; however, patients with metastatic disease who have progressed (as defined by objective response criteria for solid measurable tumor; tumor marker elevation alone is not sufficient) on a CEA-containing vaccine, may be enrolled to this study as they arise if they meet the patient eligibility criteria, but will be added-in outside of the eight established cohorts, at the currently established safe dose level; additionally, these patients will receive only the rF-CEA(6D)-TRICOM vaccine (possibly along with GM-CSF if cohort 7 is the currently established safe dose level), but otherwise will be treated according to the protocol as any other patient on study; such additional patients will not count toward study accrual, determination of primary immunologic endpoints, or the determination of the MTD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2000-11; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Immunologic response, measured by the frequency of interferon gamma-releasing T cells specific to CAP-1, an HLA-A2 restricted epitope of CEA, as measured by the ELISPOT assay | Up to 3 months after completion of study treatment
  Pre and post-vaccination CTL precursor frequencies will be calculated so that changes in CTL precursor frequencies can be compared between dose levels of the vaccine. Also, 95% confidence intervals can be calculated for the percent increases (or decreases) in CTL precursor frequencies between dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, Principal Investigator — Lombardi Comprehensive Cancer Center at Georgetown University
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia, United States